CLINICAL TRIAL: NCT05629637
Title: Feasibility and Acceptability of Mindfulness-based Resilience Training for Problematic Alcohol Use, Mental Health, and Aggression in Rural Law Enforcement Officers
Brief Title: Feasibility and Acceptability of Mindfulness-based Resilience Training for Rural Law Enforcement Officers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 090-18; 3R01AT009841-04S1 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Problem Drinking; Aggression; Stress, Psychological
MeSH Terms: conditions — Alcoholism; Aggression; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Resilience Training (MBRT) (Experimental): MBRT is an 2.5-day program combining training in standardized mindfulness practices targeting factors that facilitate resilience, cognitive-behavioral therapy (CBT), and psychoeducation. It contains experiential and didactic exercises including body scan, sitting and walking meditation, mindful movement and discussions.
  Interventions: Behavioral: Mindfulness-Based Resilience Training (MBRT)

INTERVENTIONS:
Behavioral: Mindfulness-Based Resilience Training (MBRT) — MBRT is designed to enhance resilience in the presence of acute and chronic LEO stressors. MBRT will be delivered in a hybrid format. An intensive, 22-hour in-person training will be offered, followed by 4 weekly 90-minute zoom classes. The in-person portion of the training will span 3 days: 4 hours day 1, 6 hours day 2, and 6 hours day 3. MBRT contains experiential and didactic exercises including body scan, sitting and walking meditation, mindful movement and discussions. MBRT is designed to address stressors inherent to police work, including critical incidents, job dissatisfaction, public scrutiny, and interpersonal, affective and behavioral challenges.

SUMMARY:
Rural law enforcement officers (LEOs) are exposed to unique and significant stressors, yet have access to fewer resources, compared to urban counterparts, to mitigate harmful effects of stress. This elevates risk for maladaptive coping strategies such as problematic alcohol use, mental health consequences, and aggression and excessive use of force. The proposed supplement will assess feasibility and accessibility of Mindfulness-Based Resilience Training (MBRT), with added intervention components addressing alcohol use, in under-resourced rural LEOs to ensure success in a future multisite efficacy trial assessing effects of MBRT on mental health and behavioral outcomes.

DETAILED DESCRIPTION:
The stress inherent to policing affects both officer health as well as the safety of their respective communities. The investigators current and previous research has shown that Mindfulness-Based Resilience Training (MBRT) leads to improvement in law enforcement officer (LEO) mental health and behavioral outcomes, including alcohol use and aggression. In the investigators current multisite R01 feasibility trial of MBRT, they have successfully met key feasibility and acceptability benchmarks in urban and suburban LEO samples. What is lacking is exploration of feasibility and acceptability in rural LEOs, who face unique stressors and challenges, and an integration of evidence-based preventive intervention components to directly target problematic alcohol use. Individuals living in rural communities are recognized as a target population for health disparities research. Rural LEOs experience stressors specific to rural populations such as isolation and work-role overload, yet often have fewer resources, including less access to stress management trainings and mental health care, compared to their urban and suburban counterparts. The combination of high stress coupled with low resources supporting mental health and performance may lead to increased reliance on maladaptive behaviors, such as excessive alcohol use. Indeed, LEOs have disproportionately higher rates of alcohol use, not only affecting their own health and wellbeing but also exacerbating effects of stress on aggression and excessive force in critical incidents. Preliminary evidence suggests alcohol use may be more problematic among rural, relative to urban, LEOs. The proposed supplement would support collection of data on feasibility and acceptability of MBRT in under-resourced rural LEOs to inform further adaptations to better serve this community. Additionally, the investigators propose to integrate specific elements of an evidence-based mindfulness intervention for substance use disorders to explicitly address problematic alcohol use and associated consequences among rural LEOs, enhancing effects of MBRT on officer health, and in turn reducing aggression and excessive use of force in critical incidents. Completion of supplement aims will strengthen support for a multisite trial of an intervention that holds great potential to reduce aggression and increase health and wellbeing among urban, suburban and rural LEOs and the communities they serve.

ELIGIBILITY:
Inclusion Criteria:

* be 21-65 years old,
* demonstrate English fluency,
* be a sworn, full-time, active status law enforcement officer, and
* be willing to complete assessments at multiple time points and attend intervention groups

Exclusion Criteria:

* previous participation in mindfulness-based stress reduction (MBSR), MBRT or a similar mindfulness course,
* endorse suicidal ideation, or
* unable or unwilling to give written informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Aggression | baseline, post-intervention (4 weeks), 3 month followup
  Buss-Perry Aggression Questionnaire-Short Form. Scores range from 1-5, with higher scores indicating greater aggression.
Change in Alcohol Use Negative Consequences | baseline, post-intervention (4 weeks), 3 month followup
  Patient Reported Outcome Measurement System (PROMIS) Alcohol Use Negative Consequences.Scores range from 39-77, with higher scores indicating greater alcohol use negative consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Christopher, Principal Investigator — Pacific University
Locations (1):
- Pacific University, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: No